CLINICAL TRIAL: NCT04082793
Title: Comparison of Photobiomodulation Therapy and Sonophoresis in Improving Tempomandibular Joint Mobility and Quality of Life Among Head and Neck Cancer Survivors (PBMT-S Trial): A Triple-Blind, Randomized Controlled Trial.
Brief Title: Photobiomodulation and Sonophoresis Improving Jaw Mobility and Quality of Life Among Head and Neck Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMDU/2019/02; U1111-1235-0005 (Other Grant/Funding Number: UTN by WHO international clinical Trial Registry Platform)
Record Dates: First submitted 2019-08-31; First posted 2019-09-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer; Trismus
Keywords: Electrotherapy; Photobiomodulation; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, outcome assessors and care provider will be blinded in the study. This will be a triple blinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Experimental): Low-level laser therapy will be given to the PTMB group along with mandibular mobilization and stabilization exercises
  Interventions: Combination Product: Photobiomodulation therapy with mandibular exercises; Combination Product: Sonophoresis with mandibular exercises
- Sonophoresis group (Experimental): Ultrasonic massage with diclofenac gel will be given to the sonophoresis group along with mandibular mobilization and stabilization exercises
  Interventions: Combination Product: Photobiomodulation therapy with mandibular exercises; Combination Product: Sonophoresis with mandibular exercises

INTERVENTIONS:
Combination Product: Photobiomodulation therapy with mandibular exercises — Low-level laser therapy (BMI 1005 Laser 2200) Wavelength: 658 nm Power: 100 MW Energy density: 4J/cm2 Dose administered: 4J Mode: Pulsed Site of application: Over bilateral Temporomandibular joint Number of sessions: 3 sessions/week on alternating days for 12 minutes each, for 4 weeks Mandibular mobilization exercises Side to side movement of the jaw Forward jaw movement Tongue up Goldfish exercise (Partial opening) Goldfish exercise (Full opening) Exercise duration: 6 repetitions X 2 sets X 4 times a day Mandibular Stabilization exercises Exercise duration: 5 repetitions X 3 sec. Hold X 4 times a day
  Other Names: Low-level laser therapy
Combination Product: Sonophoresis with mandibular exercises — Ultrasound (BM1-1039) Ultrasonic massage with Diclofenac gel Frequency: 1.0 MHz Mode: Continuous Intensity: 0.8 to 1.5 W/cm2
  Site of application: Over bilateral Temporomandibular joint Number of sessions: 3 sessions per week on alternating days for 8 minutes each, for 4 weeks Mandibular mobilization exercises Side to side movement Forward jaw movement Tongue up Goldfish exercise (Partial opening) Goldfish exercise (Full opening) Exercise duration: 6 repetition X 2 sets X 4 times a day Mandibular Stabilization exercises Exercise duration: 5 repetitions X 3 sec. Hold X 4 times a day
  Other Names: Ultrasonic massage with diclofenac gel

SUMMARY:
Head and neck cancer originate from the several different anatomical subsites especially the squamous cell carcinoma. This involves mainly Oropharynx, Hypopharynx, and Larynx. The common treatment approaches for HNC is radiation therapy, alone or combined with chemotherapy and surgery. In the present scenario, very little literature is available improving the QOL by physiotherapeutic measures in patients with HNC. To improve QOL, a well-designed study is needed. The study will be a two-group pretest-posttest design. The study will include patients with HNC receiving radiation or chemotherapy. One group will receive photobiomodulation therapy and another group will receive Sonophoresis. Both the group will receive Mandibular mobilization and stabilization exercises after electrotherapy. The Algometer, Digital Vernier caliper and core measure Questionnaire-C30 (QLQ-C30) will be used as an outcome measure to measure the effect of interventions between baseline and post-interventions.

DETAILED DESCRIPTION:
The trial will include two experimental groups. The study design will be two groups pretest-posttest design. The study will recruit patients with HNC receiving radiation or chemotherapy. The study will be conducted in Tertiary care teaching hospital, in the departments of Radiotherapy and physiotherapy of Maharishi Markandeshwar Hospital, Maharishi Markandeshwar Deemed to be University, Mullana, Ambala. Total of 48 patients will be recruited in the study. Patients will be randomized by block randomization method into two groups. One group will receive Photobiomodulation therapy whereas another group will receive Sonophoresis. Mandibular mobilization and stabilization exercises will be given to both groups. The intervention will be given for 4 weeks. Three sessions of photobiomodulation therapy will be given per week on alternating days for 12 minutes, whereas three sessions of sonophoresis will also be given per week on alternating days for 8 minutes. Mandibular mobilization, as well as stabilization exercises, will be advised to perform regularly continuously for 4 weeks. There will be blinding of patients who will receive the therapy, therapist who will administer the therapy, and therapist who will assess the patients, therefore, the study will follow triple blinding.Algometer for pain measurement, Digital vernier caliper for measuring mandibular mobility and Core measure Questionnaire-C30 (QLQ-C30) for measuring the quality of life in patients with head and neck cancer will be taken as outcome measures. The outcomes will be taken before giving intervention, then again after 2 weeks of interventions and again on another 2 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Clinical diagnosis of HNC undergoing chemo and radiation therapy
* Patient having joint pain and stiffness following chemo and radiation therapy
* Patients with the age group of 18 - 70 years

Exclusion Criteria:

* Patients with Mandibular reconstruction surgery
* Patients with platelet count <80,000/µl of blood and haemoglobin count <8g/dl
* Patients with cervical spine dysfunction and nerve damage
* Patients who is not willing to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Algometer | Change from baseline, 2 weeks after intervention and at the end of 4th week will be measured.
  Algometer is a digital calibrated outcome measure, measures the pain pressure threshold.
Core measure Questionnaire-C30 (QLQ-C30) | Change from baseline, 2 weeks after intervention and at the end of 4th week will be measured.
  The questionnaire are designed to measure physical, social and psychological functions of patients with cancer. The questionnaire contains physical, social, emotional and cognitive functioning multi item scales and 9 single items. These items are pain, fatigue, financial impact, appetite loss, nausea and vomiting, diarrhea, constipation, sleep disturbance and quality of life. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Time required for administration is 10 to 15 minutes.

SECONDARY OUTCOMES:
Digital Vernier calliper | Change from baseline, 2 weeks after intervention and at the end of 4th week will be measured.
  Digital Vernier calliper measures the range of motion of mandibular mobility

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, MPT, Principal Investigator — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gautam AP, Fernandes DJ, Vidyasagar MS, Maiya AG, Vadhiraja BM. Low level laser therapy for concurrent chemoradiotherapy induced oral mucositis in head and neck cancer patients - a triple blinded randomized controlled trial. Radiother Oncol. 2012 Sep;104(3):349-54. doi: 10.1016/j.radonc.2012.06.011. Epub 2012 Aug 10. PMID 22884841
- [Background] Zecha JA, Raber-Durlacher JE, Nair RG, Epstein JB, Elad S, Hamblin MR, Barasch A, Migliorati CA, Milstein DM, Genot MT, Lansaat L, van der Brink R, Arnabat-Dominguez J, van der Molen L, Jacobi I, van Diessen J, de Lange J, Smeele LE, Schubert MM, Bensadoun RJ. Low-level laser therapy/photobiomodulation in the management of side effects of chemoradiation therapy in head and neck cancer: part 2: proposed applications and treatment protocols. Support Care Cancer. 2016 Jun;24(6):2793-805. doi: 10.1007/s00520-016-3153-y. Epub 2016 Mar 17. PMID 26984249
- [Background] Shin SM, Choi JK. Effect of indomethacin phonophoresis on the relief of temporomandibular joint pain. Cranio. 1997 Oct;15(4):345-8. doi: 10.1080/08869634.1997.11746030. PMID 9481998
- [Background] Samuel SR, Maiya GA, Babu AS, Vidyasagar MS. Effect of exercise training on functional capacity & quality of life in head & neck cancer patients receiving chemoradiotherapy. Indian J Med Res. 2013 Mar;137(3):515-20. PMID 23640558
- [Background] Samuel SR, Maiya AG, Fernandes DJ, Guddattu V, Saxena PUP, Kurian JR, Lin PJ, Mustian KM. Effectiveness of exercise-based rehabilitation on functional capacity and quality of life in head and neck cancer patients receiving chemo-radiotherapy. Support Care Cancer. 2019 Oct;27(10):3913-3920. doi: 10.1007/s00520-019-04750-z. Epub 2019 Mar 27. PMID 30919154
- See also: Effectiveness of exercise-based rehabilitation on functional capacity and quality of life in head and neck cancer patients receiving chemo-radiotherapy — https://link.springer.com/article/10.1007%2Fs00520-019-04750-z